CLINICAL TRIAL: NCT07262294
Title: The Effect of Deep Breathing Added to Core Stability Exercises in the Treatment of Patients With Ankylosing Spondylitis: A Randomized Controlled Trial
Brief Title: Deep Breathing Combined With Core Stability Exercises in the Treatment of Patients With Ankylosing Spondylitis
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariam Abdel Rahman, Lecturer of Orthopaedic Physical Therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy, Beni-Suef.
Record Dates: First submitted 2025-11-15; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Breathing exercise plus Core stability exercises (Experimental): Deep Breathing exercise is a type of exercise that engage the diaphragm to enhance the respiratory function, improve lung efficiency, and induce relaxation which improve the overall health condition.
  Interventions: Other: Exercises
- Core Stability Exercises (Active Comparator): Core Stability exercises are group of exercises designed to strengthen abdominal, back, lower limbs, and pelvis muscles which enhance posture and provide stability and body control during daily activities
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Exercises

SUMMARY:
Exercise may be considered the gold standard for the management of mechanical and functional symptoms associated with patients having AS and they are considered as a safe and effective treatment for improving strength, spinal mobility, and physical fitness in general. However, there were no definite types or doses recommended over others.

Additionally, poor posture is one of the consequences of AS due to pain, loss of flexibility, and muscular weakness which may also affect respiratory function. This faulty mechanical posture of the thoracic and cervical spine may affect the pulmonary function of these patients. Therefore, the purpose of the current study is to investigate the efficacy of deep breathing exercises added to core stability exercises in the treatment of patients suffering from AS.

DETAILED DESCRIPTION:
The management of AS typically involves a multidisciplinary approach which includes both medical and physical therapy approaches, concerning the medical treatment, NSAIDs are widely used for pain relief and inflammation control in AS patients and were recommended for the management of patients having AS. The efficacy of NSAIDs has been well-documented in research studies, Disease-modifying antirheumatic Drugs (DMARDs), including sulfasalazine and methotrexate, play a crucial role in suppressing inflammation and preventing joint damage in AS patients, or biologics, such as tumor necrosis factor (TNF) inhibitors (adalimumab, etanercept, infliximab), have transformed AS treatment by specifically targeting inflammatory pathways and significantly improving symptoms and function.

Respecting the physical therapy approach plays a crucial role aims to maintaining and improving mobility, reducing pain, enhancing overall function, correcting mal-positioning, and improving patients' psychological status in patients with ankylosing spondylitis. It usually includes a combination of exercises such as Range of Motion (ROM) exercises, strengthening exercises, Cardiovascular exercises, postural training, patient education, assistive devices, Adaptations, and monitoring. Different types of exercises have been studied for managing patients having AS, however, no specific type has been recommended over others. Additionally, up to our knowledge, there were no studies has addressed the respiratory function that may be affected with patients having AS either from postural abnormalities, lack of spinal flexibility, or generalized functional limitations. Therefore, the current study aims to evaluate if deep breathing exercises as a complementary intervention would be of some value when added to core stability exercises for patients suffering from AS.

ELIGIBILITY:
Inclusion Criteria:

* Receiving the same medical treatment
* Age range between 20 and 45 years
* Includes both male and female patients
* Diagnosed with stable ankylosing spondylitis (AS) for at least 3 months
* Not engaged in any other rehabilitation programs within the last 6 months

Exclusion Criteria:

* Presence of other systemic or neurological disorders
* Any change in medication within the last 6 months

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory function | Patients will be examined after 4 to 6 weeks
  Forced vital capacity (FVC) which measure lung volume, and it reflects the capacity of the lung.
  Forced expiratory volume in 1 second (FEV1) which measure lung velocity, and it evaluate the presence of airway obstruction.
  FEV1/FVC it the index that differentiate between obstructive and restrictive lung disease.

SECONDARY OUTCOMES:
Functional exercise capacity | Patients will be examined after 4 to 6 weeks
  The physical functional performance will be assessed by a six-minute walk test (6 MWT)